CLINICAL TRIAL: NCT02971319
Title: Exploratory Phase II Study in Patients After Treatment of High Grade Brain Tumors to Assess the Technical Performance of Tc-99m Tetrofosmin for Differentiation of Recurrence Versus Radiation Necrosis
Brief Title: Technical Performance Assessment of Tc-99m Tetrofosmin for Differentiation of Recurrence vs Radiation Necrosis in Patients With Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Proactina S.A. (Other)
Collaborators: ConsulTech GmbH (Unknown); pharmtrace (Unknown); Pharmathen S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Gliomark
Record Dates: First submitted 2016-11-16; First posted 2016-11-22 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Glioma (Diagnosis)
MeSH Terms: conditions — Glioma; Disease

INTERVENTIONS:
Device: Tc-99M-Tetrofosmin SPECT
Device: F-18 FDG PET

SUMMARY:
This study aims to assess the technical performance of Tc-99m tetrofosmin SPECT as compared to F-18 FDG PET for the differentiation of radiation necrosis from glioma relapse and to obtain estimates of diagnostic accuracy for Tc-99m tetrofosmin SPECT and F-18 FDG PET in an intra-individual comparison.

ELIGIBILITY:
Inclusion Criteria:

1. confirmed high grade glioma (e.g., anaplastic astrocytoma, glioblastoma, anaplastic oligodendroglioma, or anaplastic oligoastrocytoma)
2. being in follow-up for at least 3 months after completion of radiation therapy (with or without concurrent chemotherapy)
3. inconclusive MRI results regarding the differentiation between recurrence and radiation necrosis
4. willing and able to undergo all study procedures
5. informed consent in writing (dated and signed)

Exclusion Criteria:

1. age: less than18 years
2. if female, pregnant or breast feeding (females of child-bearing potential must use adequate contraception and must have a negative pregnancy test performed within 7 days prior to inclusion into this study)
3. contraindications for Tc-99m tetrofosmin
4. contraindications for F-18 FDG
5. close affiliation with the investigational site; e.g. first-degree relative of the investigator
6. participating in another therapeutic clinical trial or has completed study participation in another therapeutic clinical trial within 5 days of enrolment into this trial
7. having been previously enrolled in this clinical trial
8. being mentally disabled
9. mental conditions rendering the subject incapable to understand the nature, scope, and consequences of the trial
10. Being clinically unstable or requiring emergency treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-09; Primary Completion 2017-11-17 (Actual); Study Completion 2017-12-17 (Actual)

PRIMARY OUTCOMES:
Technical performance of Tc-99m tetrofosmin SPECT | assessed once within 3 weeks of inclusion

CONTACTS AND LOCATIONS:
Locations (9):
- Service de Neurologie Mazarin Hôpital Pitié-Salpêtrière, Paris, France
- Hungary (8):
  - Országos Klinikai Idegtudományi Intézet (OKITI), Budapest
  - Országos Onkológiai Intézet, Budapest
  - Pozitron-Diagnosztika Ltd., Budapest
  - Scanomed Budapest, Budapest
  - Uzsoki Utcai Kórház, Budapest
  - Debreceni Egyetem Orvos- és Egészségtudományi Centrum, Debrecen
  - Scanomed Debrecen, Debrecen
  - Pécsi Tudományegyetem, Általános, Pécs